CLINICAL TRIAL: NCT00877266
Title: Ultrasound Guidance vs. Electrical Stimulation for Perineural Catheter Insertion: A Randomized, Controlled Trial
Brief Title: Ultrasound Guidance Versus Electrical Stimulation for Perineural Catheter Insertion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Brian Ilfeld, M.D., M.S./ Principal Investigator, University of California, San Diego, Department of Anesthesiology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: US vs. NS Perineural Catheter
Record Dates: First submitted 2009-04-03; First posted 2009-04-07 (Estimated); Last update posted 2009-04-07 (Estimated); Status verified 2009-04

CONDITIONS: Postoperative Pain
Keywords: catheter; ultrasound guidance; nerve stimulation; electrical stimulation; nerve block; UCSD; timed placement; surgery; Catheter Placement Time
MeSH Terms: conditions — Pain, Postoperative | interventions — Electric Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. Ultrasound (Active Comparator): Ultrasound is randomly chosen by use of a computer program. The time for catheter placement will begin with the ultrasound probe touches the patient. Patients will be asked their discomfort on a 0-10 scale (0=no discomfort and 10=worst discomfort imaginable) and will be called the next day by the research staff.
  Interventions: Procedure: perineural mepivicaine catheter placed via ultrasound or electrical stimulation
- 2. Electrical Stimulation (Active Comparator): Nerve Stimulation (electrical stimulation) is randomly chosen using a computer program. Time of placement begins when the catheter-placement first touches the patient. After catheter placement patient is asked their discomfort on a 0-10 scale (0=no discomfort and 10=worst discomfort imaginable) and called the day after surgery by the research staff.
  Interventions: Procedure: perineural mepivicaine catheter placed via ultrasound or electrical stimulation

INTERVENTIONS:
Procedure: perineural mepivicaine catheter placed via ultrasound or electrical stimulation — Patients will be randomized to one of two groups: catheter placement via ultrasound or nerve stimulation. Placement of the catheter will be timed by research staff and discomfort level asked after placement of catheter. If the catheter is not placed by the randomized method within 15 minutes, the practitioner my switch to the alternate method. Patients will be called the morning after surgery by research staff to assess discomfort levels.

SUMMARY:
This research study is to determine the relative times for perineural catheter placement with the use of ultrasound versus electrical stimulation. The perineural catheter is placed next to the nerves through which local anesthetic is placed to provide pain control following surgery. This study may determine if one method is associated with increased success rate and patient comfort.

DETAILED DESCRIPTION:
Primary Specific Aim: To determine if the relative times for perineural catheter placement with the use of ultrasound versus electrical stimulation.

Hypothesis: Compared with the use of electrical stimulation, the use of ultrasound guidance when inserting a perineural catheter is associated with a decreased time of placement.

Secondary Specific Aim: To determine if other possible benefits of perineural catheter placement associated with the use of ultrasound guidance versus electrical stimulation.

Hypothesis: Compared with the use of electrical stimulation, the use of ultrasound guidance when inserting a perineural catheter is associated with an increased surgical block success rate and catheter-placement success rate, as well as decreased patient discomfort and incidence of venous puncture.

ELIGIBILITY:
Inclusion Criteria:

* undergoing surgery with a planned perineural catheter for postoperative analgesia
* catheter in the interscalene, infraclavicular, popliteal, or femoral anatomic location
* age 18 years or older

Exclusion Criteria:

* pregnancy
* inability to communicate with the investigators and hospital staff
* incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2007-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
The primary outcome measurement will be the time of placement for a perineural catheter using either ultrasound-guided method or electrical stimulation method. | 30 minutes

SECONDARY OUTCOMES:
Pain and discomfort as assessed by a 0-10 scale (0=no pain/discomfort and 10=worst pain/discomfort imaginable) by the research coordinator. | After catheter placement and Postoperative day 1

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, M.D., M.S., Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Medical Center, San Diego, California, United States